CLINICAL TRIAL: NCT03643731
Title: Pain Relief in Patients With Chronic Low Back Pain Using HeatTens vs. Standard Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lynn Leemans, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.U.N. 143201836092
Record Dates: First submitted 2018-08-10; First posted 2018-08-23 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Chronic Low Back Pain; Movement Evoked Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeatTens (Experimental): After baseline measurements and during 4 weeks of follow up
  Composition and dosing of the device:
  HeatTens (HV-F311-E) 2 - 108 Hz (modulation), 100 microsec (pulse duration) for 30 minutes.
  Interventions: Device: HeatTens (HV-F311-E)
- Control group (No Intervention): No intervention

INTERVENTIONS:
Device: HeatTens (HV-F311-E) — Patients need to apply the device during 30 minutes.
  Arms: HeatTens

SUMMARY:
A two-armed randomized controlled clinical trial with blind assessments and a follow-up period of 4 weeks is developed. The aim of this study is to investigate the effects of the combination of heat and TENS (HeatTENS device) on pain in people with chronic low back pain. A sample of 70 patients will be recruited. Following baseline measurements, subjects will be randomly allocated to the experimental or the control group. The experimental group will be asked to use the device on a daily basis, 30 minutes per day. The control group will have no device. After 4 weeks of FU, measurements will be repeated.

DETAILED DESCRIPTION:
Drop out:

If subjects drop out, due to any kind of reason, a new participant will be included in order to obtain the predetermined number of participants. Data collected from the participant that dropped out will be deleted and not taken into account in the further analysis.

Analysis of the samples:

Sample size is based on data from (Dailey et al. 2013). Researchers found a significant difference in the reduction of movement-evoked pain (pain during the 6 minutes' walk test (6MWT)) ((4.0 ± 2.5) on a 0-10 VAS) when compared to no TENS (5.0 ± 2.6) (p<0.05) in patients with primary fibromyalgia.

In this study the response within each subject group was normally distributed. If the true difference in the experimental and control means is 1.0, effect size is calculated to be 0,2 (by means of G*Power version 3.1.9.3). 29 experimental subjects and 29 control subjects need to be included to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. To take into account a 15% loss of data sample size is inflated up to 33 per group (n/0.85). Sample size is augmented by 10% per potential confounding factor (i.e. age and sex). The total sample size to be recruited will be 70 subjects.

Statistical analysis:

The person to conduct the statistical analyses will be Lynn Leemans (Human Physiology and Anatomy (KIMA), Vrije Universiteit Brussel).

An intention-to-treat analysis will be performed so that the integrity of the randomization is ensured. Normality will be checked via the Shapiro-Wilk test.

To ensure good balance of participant characteristics in each group at baseline, stratification is used. Changes in differences between both treatment groups after the intervention period (at 4w) will be analyzed using repeated measures ANOVA for the following variables: sensitivity to movement-evoked pain, quality of life, pressure pain thresholds, temporal summation and conditioned pain modulation.

If the modulus of the partial correlation of potential confounding factors age and sex with the primary outcome values equals minimum 0.3, these covariates of prognostic values will be added as covariates in the ANOVA model.

As a secondary analysis, a linear regression analysis will be used with the following dependent factors: BMI, and as independent factors: sensitivity to movement-evoked pain, pressure pain thresholds, temporal summation, conditioned pain modulation, fear avoidance beliefs and quality of life.

Significance value for all tests will be set at p < 0.05. All analyses will be performed using SPSS 20 for Mac.

Quality control and quality assurance:

All electronic data will be stored on the shared drive of a university computer, which is encrypted; and on a password protected laptop belonging to the principal researcher (Lynn Leemans). Transfer of data will only be done if essential.

All anonymised data will be stored for up to four years to allow for access before publication, and may be required at a later date for further analysis and auditing. All personal data, including health questionnaires and signed consent forms, will be destroyed within 12 months of the study finishing.

Publication policy:

Both parties (VUB and Omron) acknowledge the importance of public disclosure of information collected of generated because of this clinical study. Omron retains the ability before publication to verify and ensure correct and accurate information is represented of the product and the brand used (product names, product types, brand name, product code) with no influence of the scientific results and conclusions of the integrity of the publication.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific LBP for at least 3 months' duration: non-specific LBP implies that patients are not allowed to have any evidence of specific spinal pathology (e.g., hernia, spinal stenosis, spondylolisthesis, infection, spinal fracture or malignancy).

Exclusion Criteria:

* spinal surgery in the past 6 months
* severe underlying comorbidity (like diagnosed diabetes, cardiovascular problems, etc.),
* pregnant or given birth in the preceding year,
* having initiated a new LBP treatment in the 6 weeks prior to study participation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Movement Evoked Pain | Change from Baseline Movement Evoked Pain after treatment and at 4 weeks
  Pain that is experienced in response to a physical task. Participants will perform 5 physical tasks (= 1) grasping toes with fingertips in a sitting position; 2) forward bending from standing; 3) picking up paper from standing; 4) long-sitting from supine and 5) lifting a 5kg box from floor to table). Participants will provide a pain rating on a 11 points Numeric Rating Scale (NRS) with the endpoints no pain" (0) and "excruciating pain" (10)

SECONDARY OUTCOMES:
5 minute walk test (5MWT) | Change from Baseline 5MWT after treatment and at 4 weeks
  Subjects need to walk as far as possible in 5 minutes
Pressure Pain Threshold (PPT) | Change from Baseline Pressure Pain Threshold after treatment and at 4 weeks
  This measures deep tissue hyperalgesia, defined as the point at witch the pressure sensation turned into pain.
Temporal summation (TS) | Change from Baseline Tempral Summation after treatment and at 4 weeks
  This is used to evaluate (endogenous) pain facilitation. Temporal summation is induced trough 10 pressure pulses with a hand held algemener (Somedic AB, Farsta, Sweden) at the Pressure Pain Threshold intensity. Patients will rate their pain level at the first, 5th and 10th pulse. Participants will provide a pain rating on a 11 points Numeric Rating Scale (NRS) with the endpoints no pain" (0) and "excruciating pain" (10)
Conditioned pain modulation | Change from Baseline Conditioned pain modulation after treatment and at 4 weeks
  This is used to evaluate the ability of the brain to moderate pain. In Conditioned pain modulation, a painful stimulus produces a decrease in pain outside the area of the applied stimulus. The mechanism behind it can be described as "pain inhibits pain". To induce pain and therefore trigger CPM response, participants put their hand in cold water for 2 minutes. Patients need to rate their level of pain (applied stimulus) on a 11 points Numeric Rating Scale (NRS) with the endpoints no pain" (0) and "excruciating pain" (10)
Fear Avoidance Beliefs Questionnaire- work | Change from Baseline Fear Avoidance Beliefs Questionnaire after treatment and at 4 weeks
  Catastrophic thoughts and believes in chronic pain patients
Quality of life (SF-36) | Change from Baseline Quality of Life after treatment and at 4 weeks
  Quality of life, due to their low back pain, experienced by the patients will be evaluated
Central sensitization inventory | Change from Baseline Central sensitization inventory after treatment and at 4 weeks
  To report signs of central sensitization and its overlapping symptoms
Body composition and Body Mass Index (BMI) | Change from Baseline Body composition and BMI at 4 weeks follow up
  These two assessments are used to evaluate overweight and obesity in chronic low back patients. Body composition will be described in percentages of fat and muscle (%). Weight (in kilograms) and height (in meters) will be assessed as well and will be combined to report BMI in kg/m^2. The ViVa body composition monitor (OMRON) will be used for these measurements. Accepted classification for overweight and obesity by BMI: <18.5 = underweight; 18.5-24.5 = normal; 25.0-29.9 = overweight and >30.0= obesity.

CONTACTS AND LOCATIONS:
Overall Officials: David Beckwée, PhD, Study Director
Locations (1):
- Vrije Universiteit Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leemans L, Elma O, Nijs J, Wideman TH, Siffain C, den Bandt H, Van Laere S, Beckwee D. Transcutaneous electrical nerve stimulation and heat to reduce pain in a chronic low back pain population: a randomized controlled clinical trial. Braz J Phys Ther. 2021 Jan-Feb;25(1):86-96. doi: 10.1016/j.bjpt.2020.04.001. Epub 2020 May 12. PMID 32434666